CLINICAL TRIAL: NCT04352465
Title: Treatment of Acute Respiratory Syndrome Resulting From the Inflammatory Process of COVID-19 Infection Using Methotrexate-loaded Nanoparticles: A Phase I/II Study
Brief Title: Efficacy and Safety of MTX-loaded Nanoparticles to Treat Severe COVID-19 Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: InCor Heart Institute (Other); Hospital Santa Marcelina (Other); Prevent Senior Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LDE-MTX_COVID19
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: The study will be divided in 3 phases:
  Phase A: subjects will be dosed 20 mg of MTX IV, once per week (total of 4 doses).
  Phase B: will only start after 2nd or 3rd administration of phase A. Subjects will be dosed 30 mg of MTX IV, once per week (total of 4 doses).
  Phase C: will only start after 2nd or 3rd administration of phase B. Subjects will be dosed 40 mg of MTX IV, once per week (total of 4 doses).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Phase A: subjects will be dosed 20 mg of MTX IV, once per week (total of 4 doses).
  Interventions: Drug: Methotrexate
- B (Experimental): Phase B: will only start after 2nd or 3rd administration of phase A. Subjects will be dosed 30 mg of MTX IV, once per week (total of 4 doses).
  Interventions: Drug: Methotrexate
- C (Experimental): Phase C: will only start after 2nd or 3rd administration of phase B. Subjects will be dosed 40 mg of MTX IV, once per week (total of 4 doses).
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Phase A: Subjects will be dosed 20 mg of MTX IV, once per week (total of 4 doses).
  Other Names: MTX-loaded nanoparticles
  Arms: A
Drug: Methotrexate — Phase B: Subjects will be dosed 30 mg of MTX IV, once per week (total of 4 doses).
  Other Names: MTX-loaded nanoparticles
  Arms: B
Drug: Methotrexate — Phase C: Subjects will be dosed 40 mg of MTX IV, once per week (total of 4 doses).
  Other Names: MTX-loaded nanoparticles
  Arms: C

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of MTX-loaded nanoparticles in three different doses to treat severe COVID-19 patients.

DETAILED DESCRIPTION:
Patients with acute lung injury caused by COVID-19 disease are experiencing an inflammatory reaction that can be harmful and worsen the severity of the clinical condition. Thus, the use of MTX-loaded nanoparticules in patients with acute lung injury secondary to COVID-19 aims to decrease the exacerbated inflammatory reaction leading to a decrease in cell damage caused by this inflammatory process in patients.

The study will be divided in 3 phases:

Phase A (n=4): IV administration of 20 mg of MTX-loaded nanoparticles. Four doses of Investigational Product (IP) will be administered, once per week. If patients show clinical improvement after 2nd or 3rd administration, the next phase will start.

Phase B (n=12): IV administration of 30 mg of MTX-loaded nanoparticles. Four doses of Investigational Product (IP) will be administered, once per week. If patients show clinical improvement after 2nd or 3rd administration, the next phase will start.

Fase C (n=26): IV administration of 40 mg of MTX-loaded nanoparticules. Four doses of Investigational Product (IP) will be administered, once per week.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or legal representative.
2. Male or female, aged ≥ 18 years;
3. Acute respiratory distress syndrome; with imminent risk of death, and with chest CT scan with pulmonary impairment greater than 50%;
4. Confirmed or pending diagnosis of COVID-19.

Exclusion Criteria:

1. Pleural effusion > 150mL or ascites > 200mL;
2. Chronic liver disease;
3. ALT and AST serum levels >= three times the upper limit of normality;
4. Renal failure (dialysis)
5. Multiple organ failure

7. Concomitant use or use in the last 7 days of cell therapy with stem cells; 8. Any clinical or laboratory condition or comorbidity that, at medical discretion, 9. Known hypersensitivity to the investigational product; 10. Subject who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinical conditions | 21 days
  Clinical condition will be measured by lung injuries

SECONDARY OUTCOMES:
Change of Clinical symptoms - respiratory rate | 21 days
  Evaluation of Pneumonia change
Hypoxia | 21 days
  oxygen saturation
Changes of blood oxygen | 21 days
  PaO2 / FiO2 ratio
Inflammatory parameters | 21 days
  C-reactive protein and ferritin
Evolution of Acute Respiratory Syndrome | 21 days
  Time to wean off oxygen invasive ventilatory support
Hospital discharge | 21 dyas
  Time to be discharged from hospital
ICU discharge | 21 days
  Time to be discharged from ICU
Rate of mortality | 4 months
  Evaluation of change in acute respiratory syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Prevent Senior Private Operadora de Saúde LTDA., São Paulo, Brazil